CLINICAL TRIAL: NCT03488849
Title: SureCRIC Standardized Patient Study
Status: Completed | Type: Interventional
Sponsor: InnoVital Systems, Inc. (Industry)
Collaborators: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SureCRIC_SP1; W81XWH-14-C-0011 (Other: Defense Health Program)
Record Dates: First submitted 2018-03-23; First posted 2018-04-05 (Actual); Results first posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-10

CONDITIONS: Airway Obstruction
Keywords: cricothyrotomy
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Intervention Model Description: The study is a two-arm, open-label study involving users - largely licensed paramedics or combat medics - identifying the cricothyroid membranes on healthy volunteers. The Control Group will perform cricothyroid membrane identification on healthy male and female volunteers of varying heights, weights, and BMI's with the standard, freehand approach. The Experimental Group will perform cricothyroid membrane identification on the volunteers with the help of the SureCRIC.
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (2):
- SureCRIC (Experimental): SureCRIC-aided cricothyroid membrane identification
  Interventions: Device: SureCRIC
- Freehand (Active Comparator): Freehand cricothyroid membrane identification
  Interventions: Other: Freehand

INTERVENTIONS:
Device: SureCRIC — SureCRIC is intended to be used as an accessory to cricothyrotomy and tracheotomy devices, helping to identify and stabilize anatomical landmarks for establishing an airway.
  Arms: SureCRIC
Other: Freehand — Freehand palpation approach to identification of the cricothyroid membrane
  Arms: Freehand

SUMMARY:
SureCRIC is intended to be used as an accessory to cricothyrotomy and tracheotomy devices, helping to identify and stabilize anatomical landmarks for establishing an airway.

Cricothyroid membrane identification accuracy has been reported to be 30-62% in the literature [Bai15, Ell10, Kri15, Lam15]. The current study assesses SureCRIC-assisted medic performance in identifying the cricothyroid membrane in a diverse standardized patient population.

DETAILED DESCRIPTION:
The study is a two-arm, open-label study involving users - largely licensed paramedics or combat medics - identifying the cricothyroid membranes on healthy volunteers. The Control Group will perform cricothyroid membrane identification on healthy male and female volunteers of varying heights, weights, and BMI's with the standard, freehand approach. The Experimental Group will perform cricothyroid membrane identification on the volunteers with the help of the SureCRIC. An expert verifier (senior otolaryngologist) will verify correct cricothyroid membrane identification and will not be blinded in order to reduce any error that may be introduced by SureCRIC removal and subsequent skin movement. The primary endpoint is a pass/fail assessment for cricothyroid membrane identification. The main secondary endpoint is time to cricothyroid membrane identification. The study design was recommended by FDA. The study, per FDA guidance, is not designed for statistical comparisons and only descriptive statistics are provided.

ELIGIBILITY:
Participants (Users):

Inclusion Criteria:

* Paramedic or military combat medic
* Trained to perform a cricothyrotomy

Exclusion Criteria:

* Current or former instructor of cricothyrotomy, airway management, or anatomy
* Experience performing cricothyrotomy on a patient in the last 6 months
* Training on cricothyrotomy in the last 3 months
* Previous or current participation in a study related to cricothyrotomy
* Any condition or physical impairment that limits dexterity and/or tactile feedback
* Performed two or more cricothyrotomies on live humans
* Previous exposure to the SureCRIC

Healthy Volunteers (Standardized Patients):

Inclusion Criteria:

* Less than 10th percentile height female
* 50th percentile height female
* Greater than 90th percentile height female
* Less than 10th percentile height male
* 50th percentile height male
* Greater than 90th percentile height male

Exclusion Criteria:

* Previous exposure to the SureCRIC
* Age under 18 or over 60
* Any skin condition including, but not limited to, eczema and hives
* Skin that is thin, fragile, sensitive and/or prone to redness or irritation including skin that maintains a red, irritated appearance after the light application of pressure
* Easy bruising or use of any blood thinning medication (including aspirin)
* Beard on the neck
* Use of a steroid medication by mouth or in a topical formulation like a cream or ointment
* Any of the following chronic conditions: chronic kidney disease, chronic liver disease, coagulation disorders such as hemophilia or von Willebrand disease, low or dysfunctional platelets (e.g., thrombocytopenia), leukemia, Cushing's syndrome, Ehlers Danlos syndrome, celiac disease, any condition that causes easy bruising or sensitive or fragile skin.
* Previous neck surgery, previous neck trauma, thyroid mass or enlargement, or other neck abnormalities
* Any condition that would make lying supine or without a pillow painful or impossible

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Center for Human Factors in Healthcare, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bair AE, Chima R. The inaccuracy of using landmark techniques for cricothyroid membrane identification: a comparison of three techniques. Acad Emerg Med. 2015 Aug;22(8):908-14. doi: 10.1111/acem.12732. Epub 2015 Jul 21. PMID 26198864
- [Background] Elliott DS, Baker PA, Scott MR, Birch CW, Thompson JM. Accuracy of surface landmark identification for cannula cricothyroidotomy. Anaesthesia. 2010 Sep;65(9):889-94. doi: 10.1111/j.1365-2044.2010.06425.x. PMID 20645953
- [Background] Kristensen MS, Teoh WH, Rudolph SS, Tvede MF, Hesselfeldt R, Borglum J, Lohse T, Hansen LN. Structured approach to ultrasound-guided identification of the cricothyroid membrane: a randomized comparison with the palpation method in the morbidly obese. Br J Anaesth. 2015 Jun;114(6):1003-4. doi: 10.1093/bja/aev123. No abstract available. PMID 25991744
- [Background] Lamb A, Zhang J, Hung O, Flemming B, Mullen T, Bissell MB, Arseneau I. Accuracy of identifying the cricothyroid membrane by anesthesia trainees and staff in a Canadian institution. Can J Anaesth. 2015 May;62(5):495-503. doi: 10.1007/s12630-015-0326-y. Epub 2015 Jan 31. PMID 25637060

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We aimed to include 2 groups of 10 participants. One group for the SureCRIC arm and one group for the freehand arm. 12 participants/group were recruited to fill this quota. Ultimately, 10 participants were included in the SureCRIC arm and 8 in the freehand arm due to no-shows/cancellations. The 18 participants represented novice target end users: paramedics & military medics. Each of the 18 participants tested on 6 healthy standardized patients: M's & F's of <10th, 50th & >90th %ile heights.
Groups:
- Standardized Patients: Healthy males and females representing the <10th, 50th and >90th percentile heights.
Period: Overall Study
Arm/Group | SureCRIC | Freehand | Standardized Patients
Started | 10 | 8 | 6
Completed | 10 | 8 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants: Exposure to human cadaver practice (10% of SureCRIC participants vs. 50% of freehand participants); real-world procedural performance (0% of SureCRIC participants vs. 37.5% of freehand participants).
  Standardized Patients: Healthy volunteers.
Groups:
- Standardized Patients: Healthy male and female volunteers corresponding to the 5th, 50th and 95th percentile heights.
- Total: Total of all reporting groups
Arm/Group | SureCRIC | Freehand | Standardized Patients | Total
Number analyzed (Participants) | 10 | 8 | 6 | 24
Age, Customized [Count of Participants; unit: Participants]
  Between 18-65 | 10 | 8 | 6 | 24
Sex/Gender, Customized [Count of Participants; unit: Participants]
  M or F (not recorded) | 10 | 8 | 0 | 18
  male | 0 | 0 | 3 | 3
  female | 0 | 0 | 3 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
First-hand, real-world human performance [Count of Participants; unit: Participants] | 0 | 3 | 0 | 3
Human cadaver training [Count of Participants; unit: Participants] | 1 | 4 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Paramedics/Combat Medics Who Accurately Identified the Cricothyroid Membrane on Standardized Patients of Different Sizes
Description: pass/fail assessment for CTM identification as gauged by expert (senior orolaryngologist)
Time Frame: 1 day
Population: paramedic or combat medic identified cricothyroid membranes on standardized patients as judged by an expert otolaryngologist
Measure: Count of Participants; unit: Participants
Groups:
- Standardized Patient: Healthy volunteers - males and females corresponding to the 5th, 50th, and 95th percentile heights
Arm/Group | SureCRIC | Freehand | Standardized Patient
Number analyzed (Participants) | 10 | 8 | 6
Participants
  CTM Identification Success in Less than 10th Percentile Height Female Standardized Patient | 6 | 7 | NA — participants are identifying the cricothyroid membrane on the standardized patient
  CTM Identification Success in 50th Percentile Height Female Standardized Patient | 8 | 5 | NA — participants are identifying the cricothyroid membrane on the standardized patient
  CTM Identification Success in Greater than 90th Percentile Height Female Standardized Patient | 10 | 7 | NA — participants are identifying the cricothyroid membrane on the standardized patient
  CTM Identification Success in Less than 10th Percentile Male Height Standardized Patient | 9 | 7 | NA — participants are identifying the cricothyroid membrane on the standardized patient
  CTM Identification Success in 50th Percentile Male Height Standardized Patient | 8 | 4 | NA — participants are identifying the cricothyroid membrane on the standardized patient
  CTM Identification Success in Greater than 90th Percentile Male Height Standardized Patient | 9 | 7 | NA — participants are identifying the cricothyroid membrane on the standardized patient

2. Secondary Outcome: Time to Cricothyroid Membrane Identification
Description: time to cricothyroid membrane identification as measured by direct observation
Time Frame: 1 day
Population: paramedic or combat medic
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | SureCRIC | Freehand
Number analyzed (Participants) | 10 | 8
seconds | 34.4 (13.4) | 10 (7.6)

ADVERSE EVENTS:
Time Frame: 1day
Description: standardized patient bruising, injury
Groups:
- Standardized Patients: Healthy volunteers corresponding to the <10th, 50th and >90th percentile heights.
Arm/Group | SureCRIC | Freehand | Standardized Patients
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SureCRIC (N=10) | Freehand (N=8) | Standardized Patients (N=6)
injury including bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) — injury from tools, devices, palpation etc. to either the participant (paramedic/combat medic) or standardized patient

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT03488849/Prot_SAP_001.pdf